CLINICAL TRIAL: NCT04614688
Title: Assessing the Impact of a Patient Education Platform to Augment the Informed Consent Process for Obstetrics and Gynecology Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-215
Record Dates: First submitted 2020-10-19; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Hysteroscopy Surgery; Informed Consent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Education Group (Experimental): Patients in this group will undergo the standard physician-led informed consent process and then be provided with an interactive patient education platform for hysteroscopy on a tablet available in the clinic for up to one hour of time. After the patient has explored the patient education platform, they will be given a post-consent survey which will measure their understanding of the surgery, their readiness for the surgery, and their satisfaction with the consent process.
  Interventions: Behavioral: Patient Education Platform
- Standard Consent Group (No Intervention): Patients in this group will undergo the standard physician-led informed consent process only. After they have consented to the surgery, they will be given a post-consent survey which will measure their understanding of the surgery, their readiness for the surgery, and their satisfaction with the consent process.

INTERVENTIONS:
Behavioral: Patient Education Platform — The patient education platform for hysteroscopy surgery is a website platform which has patient education materials regarding hysteroscopy procedures in the format of pictures, videos, and text. Information on this platform includes anatomy of the surgery area, what to expect, reasons for the surgery, ways to prepare for the surgery, and recovering from the surgery.
  Arms: Patient Education Group

SUMMARY:
Over the past few decades, there has been a shift in the informed consent process, whereby the focus is centered on patient comprehension, preparedness and satisfaction. When comparing interactive informed consent processes, such as the use of educational pathways, videos, written communication, and the traditional conversational based process, the results are conflicting. Some studies report improved patient comprehension, satisfaction and preparedness with the informed consent interventions, while others found no difference. The purpose of this study is to determine whether the use of a preoperative interactive patient education pathway improves patient comprehension, preparedness and satisfaction prior to undergoing a hysteroscopic procedure.

DETAILED DESCRIPTION:
Informed consent is dependent on three criteria; the patient must be competent, relevant information including risks, benefits and alternatives must be clearly communicated, and the acceptance of treatment must be voluntary. The consent process usually occurs in the office setting through physician-led verbal communication. Despite satisfying the three criteria of informed consent, many patients leave the office with an inadequate understanding of the treatment they have consented to.

The purpose of this study is to use an interactive patient education pathway as an adjunct to the informed consent process for patients undergoing hysteroscopy. This will be done using a randomized controlled trial design.

Patients will be randomized to the control group (standard consent process) or the education group (standard consent process augmented by access to an interactive hysteroscopy teaching platform).

All patients will undergo the standard physician-led informed consent process. Patients from both groups will be asked to complete a post-informed consent questionnaire to assess their understanding of their upcoming procedure, preparedness for the procedure, and satisfaction with the informed consent process, be that through the traditional method or the interactive patient education portal.

ELIGIBILITY:
Inclusion Criteria:

* Women planning on undergoing a hysteroscopy procedure

Exclusion Criteria:

* Women NOT planning on undergoing a hysteroscopy procedure

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Patient Comprehension of their Upcoming Surgery | After (but same day as) the patient has consented to surgery (control group) or after (but same day as) the patient has consented to surgery and explored the patient education platform (experimental group).
  Patient comprehension of their upcoming surgery will be measured using a survey given after the patient has consented to their surgery (control group) and after viewing the patient education platform (experimental group). The survey will ask the patient to name a benefit, risk, discomfort, and indication of the procedure, as well as a consequence to not having the procedure. One point will be given for each correct answer. Comprehension will be measured using a mean.

SECONDARY OUTCOMES:
Patient Preparedness for their Upcoming Surgery | After (but same day as) the patient has consented to surgery (control group) or after (but same day as) the patient has consented to surgery and explored the patient education platform (experimental group).
  Patient preparedness for the upcoming surgery will be measured using a survey given after the patient has consented to their surgery (control group) and after viewing the patient education platform (experimental group). Patients will be asked to indicate how prepared they feel on a 5-point Likert scale with 1 = Very Prepared and 5 = Very Unprepared.
Patient Satisfaction with the Consent Process | After (but same day as) the patient has consented to surgery (control group) or after (but same day as) the patient has consented to surgery and explored the patient education platform (experimental group).
  Satisfaction with the consent process will be measured using a survey given after the patient has consented to their surgery (control group) and after viewing the patient education platform (experimental group). Patients will be asked how much time they think was spent on the consent process (vs. actual time spent, measured using a stop watch). Difference between perceived time and actual time will be calculated. Patients will also be asked if certain aspects of the consent process were covered by the doctor during the discussion (e.g. "Was the procedure explained to you?", "Were the risks explained to you?"). Answer options will be "Yes/No". Patients will be asked if they received enough information to make a sound decision and if their questions were answered to their satisfaction. Answer options will be "Yes/No" Patient satisfaction will be determined using frequency counts.

CONTACTS AND LOCATIONS:
Overall Officials: Eliane Shore, MD, Principal Investigator — Unity Health Toronto